CLINICAL TRIAL: NCT00190255
Title: Pharmacogenetics of Gastrointestinal Bleeding Under Nonsteroidal Anti-inflammatory Drugs : the Role of Cytochrome P450 2C9
Brief Title: Pharmacogenetics of Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department Clinical Research of developpement
Other Study IDs: P030412
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2007-03

CONDITIONS: Gastrointestinal Hemorrhage; Stomach Ulcer; Non-steroidal Anti-inflammatory Drug Sensitivity
Keywords: gastrointestinal haemorrhage; stomach ulcer; anti-inflammatory agents, non-steroidal; CYP2C9 protein, human; genotype; pharmacogenetics
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Stomach Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastrointestinal bleeding is a severe adverse effect occurring in subjects secondary to the use of nonsteroidal anti-inflammatory drugs (NSAIDs). The enzyme CYP2C9 is responsible for the elimination of several NSAIDs. This protein is inactive in 12% of the subjects because of genetic mutations. We hypothesized that individuals carrying such mutations should be at higher risk of gastrointestinal bleeding since they display decreased NSAIDs elimination.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: CY2PC9 genotyping — CY2PC9 genotyping

SUMMARY:
Gastrointestinal bleeding is a severe adverse effect occurring in subjects secondary to the use of nonsteroidal anti-inflammatory drugs (NSAIDs). The enzyme CYP2C9 is responsible for the elimination of several NSAIDs. This protein is inactive in 12% of the subjects because of genetic mutations. We hypothesized that individuals carrying such mutations should be at higher risk of gastrointestinal bleeding since they display decreased NSAIDs elimination.

DETAILED DESCRIPTION:
Gastrointestinal bleeding is a severe adverse effect occurring in subjects secondary to the use of nonsteroidal anti-inflammatory drugs (NSAIDs). The enzyme CYP2C9 is responsible for the elimination of most NSAIDs. Several polymorphisms have been observed in CYP2C9. Of these, the CYP2C9*3 allele, found in 12% of caucasian subjects, leads to reduced function of the enzyme.

We hypothesized that individuals carrying this mutation should be at higher risk of gastrointestinal bleeding since they display decreased elimination of some NSAIDs.

The purpose of this study is to determine whether the frequency for CYP2C9*3 variant allele is increased in subjects using NSAIDs metabolized by CYP2C9 in comparison with subjects under NSAIDs not metabolized by this enzyme.

The study groups consist of 200 patients suffering from gastrointestinal bleeding after NSAIDs use, divided in 100 patients using NSAIDs metabolized by CYP2C9 and 100 patients using other NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Upper gastrointestinal bleeding revealed by hematemesis, melena or lowering of at least 2g/dl of haemoglobin
* Endoscopic report of gastrointestinal ulcer or haemorrhagic lesion
* Immediate antecedents of NSAID therapy

Exclusion Criteria:

* Cirrhosis (Child B or C)
* Coma
* Concomitant therapy with substrates or inhibitors of CYP2C9 : ketoconazole, itraconazole, ritonavir, phenobarbital, rifampicin, depakine, phenytoin, St John's worts
* Patients treated by a NSAID metabolized by CYP2C9 and a NSAID not metabolized by CYP2C9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Upper gastrointestinal bleeding revealed by hematemesis, melena or lowering of at least 2g/dl of haemoglobin
  * Endoscopic report of gastrointestinal ulcer or haemorrhagic lesion
  * Immediate antecedents of NSAID therapy
  Exclusion Criteria:
  * Cirrhosis (Child B or C)
  * Coma
  * Concomitant therapy with substrates or inhibitors of CYP2C9 : ketoconazole, itraconazole, ritonavir, phenobarbital, rifampicin, depakine, phenytoin, St John's worts
  * Patients treated by a NSAID metabolized by CYP2C9 and a NSAID not metabolized by CYP2C9
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CARBONNELL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Laurent BECQUEMONT, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Service d'hépato-gastroentérologie, Hôpital Saint Antoine, Paris
  - Service d'hépato-gastroentérologie, Hôpital Pitié Salpétrière, Paris
  - : Service d'hépato-gastroentérologie, Hôpital Henri Mondor, Paris
  - Service d'hépato-gastroentérologie, Hôpital Paul BROUSSE, Villejuif

REFERENCES:
- [Background] Martin JH, Begg EJ, Kennedy MA, Roberts R, Barclay ML. Is cytochrome P450 2C9 genotype associated with NSAID gastric ulceration? Br J Clin Pharmacol. 2001 Jun;51(6):627-30. doi: 10.1046/j.0306-5251.2001.01398.x. PMID 11422024
- [Background] Martinez C, Blanco G, Ladero JM, Garcia-Martin E, Taxonera C, Gamito FG, Diaz-Rubio M, Agundez JA. Genetic predisposition to acute gastrointestinal bleeding after NSAIDs use. Br J Pharmacol. 2004 Jan;141(2):205-8. doi: 10.1038/sj.bjp.0705623. Epub 2004 Jan 5. PMID 14707031